CLINICAL TRIAL: NCT06919458
Title: Seven Day Versus Fourteen-day Corticosteroid in Patients With Severe Alcohol -Associated Hepatitis- A Double Blind Randomized Controlled Trail (STASH II)
Brief Title: Short Course Steroids in Alcohol Associated Hepatitis
Acronym: STASHII
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Collaborators: Mahatma Gandhi Medical College (Other); Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Kalinga Institute of Medical Sciences, Bhubaneswar (Unknown); Apollo Gleneagles Hospitals, Kolkata (Other)
Responsible Party: Principal Investigator, Anand Kulkarni, Dr, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAAH-01; CTRI/2025/03/083463 (Registry Identifier: Clinical Trial Registry-India)
Record Dates: First submitted 2025-04-02; First posted 2025-04-09 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Alcoholic Hepatitis
Keywords: STASH II; corticosteroids; infections
MeSH Terms: conditions — Hepatitis, Alcoholic; Infections | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: ID specialist will be blinded to the trial group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisolone dose of 40mg/day for 7 days (Active Comparator): Participants satisfying the inclusion criteria will be randomly allocated. Participants in Group A will receive prednisolone dose of 40 mg/day for 7 days after which the participants will recieve seven days of prednisolone 40 mg/day for next 7 days provided they had responded on day 7 based on Lille score
  Interventions: Drug: Prednisolone 40 mg
- Prednisolone dose of 40mg/day for 14 days (Active Comparator): Participants satisfying the inclusion criteria will be randomly allocated. Participants in Group B will receive prednisolone dose of 40 mg/day for 14 days only if they respond to on day 7 based on Lille score
  Interventions: Drug: Prednisolone 40 mg

INTERVENTIONS:
Drug: Prednisolone 40 mg — Patients will be screened for infection till 90 days from the day of initiation of prednisolone. the three patient arms will be compared for severity scores of the disease, rate and severity of infections, diabetic control, post-treatment outcomes, and mortality.

SUMMARY:
Alcohol-associated hepatitis (AAH) is one of the most severe manifestations of the spectrum of alcohol related liver disease (ARLD), with high morbidity and mortality. Currently, corticosteroids are the standard of care for patients with severe AAH, but no consensus exists on the dosing schedule of steroids. The investigators have recently demonstrated that tapering prednisolone over 4 weeks reduces the risk of infections at day 90. However, the investigators wanted to test whether the reduction in the duration of therapy would provide a similar benefit as tapering the dose of prednisolone. Therefore, the investigators planned to assess the impact of a shorter duration of prednisolone on outcomes, including the incidence of infections, survival and adverse events. One group will receive 7 days of prednisolone followed by a placebo for the next seven days, and the other group will receive 40 mg of prednisolone for 14 days. Prednisolone will be stopped in case of non-response and/or adverse events to the drug. All infections will be diagnosed by an ID specialist who is blind to the allocated group.

DETAILED DESCRIPTION:
Alcohol-associated hepatitis (AAH) is one of the most severe manifestations of the spectrum of alcohol-related liver disease (ARLD). Severe alcohol-associated hepatitis (AAH), defined by a Maddrey's Discriminant Function score (mDF) greater than 32, can be associated with a greater than 20-30% mortality rate within 3 months in patients.1 Several therapies have been evaluated for AAH, but only corticosteroids and pentoxifylline have shown some benefit in the treatment.2 Currently, corticosteroids (prednisolone 40 mg or equivalent dose) are the recommended standard of care for patients with AAH who have severe disease identified by NIAAA criteria as steroids short-term mortality benefits.3 However, the dosing schedule of corticosteroids is not clearly stated. American Association for the Study of Liver Disease (AASLD), the European Association for the Study of Liver (EASL), and the American College of Gastroenterology (ACG) recommend using a daily dose of 40mg of oral prednisolone for 28 days, followed by abrupt discontinuation.4-6 While EASL mentions tapering doses over 2 to 3 weeks after 40 mg of therapy for 4 weeks or abrupt withdrawal. (Table 1) The reason for this dosing schedule of 40 mg for 4 weeks has been derived from studies performed more than 4 decades ago.7,8 The investigators recently reported that tapering of prednisolone over 4 weeks reduces the risk of infection in these patients compared to those receiving fixed 40 mg dose of prednisolone. The average daily prednisolone dose was 40 mg/day in the fixed-dose group compared with only 28.4±6.1 mg/day in the tapered-dose group (P<0.001), although the duration of prednisolone therapy was similar in both groups (22.1±9.1 days in the fixed-dose arm vs. 23±8.8 days in the tapered-dose arm; P=0.44). The lower dose of prednisolone led to a reduction in the incidence of infections. To continue the research in this area, the investigators wanted to test whether reducing the duration of prednisolone reduces infections.

- All patients of AAH with MELD score >21 and/or mDF >32 visiting the hospital (OPD/IPD) in the study period who do not have any contraindications for oral prednisolone therapy will be included in the study.

This is a double-blinded RCT. The CTC will generate a random allocation sequence using computer-based random numbers. Treatment allocation will be performed using block randomization with a block size of 10. The CTC will randomly assign patients to either the prednisolone 7-day or 14-day prednisolone using the sealed opaque sequentially numbered envelopes (SNOSE) method. The patients and investigators will be blinded to the allocated treatment. The drugs will be administered by the CTC.

STUDY METHODS / STUDY PROCEDURE / METHODS OF ASSESSMENT - All patients with AAH will be screened for inclusion in the study. Investigations to exclude infections before initiation of corticosteroids, including complete blood counts, cultures (blood, ascitic and urine), serum procalcitonin levels and Chest radiographs, will be performed. Design of infection screening is based on previous studies (8,9,10). Randomisation will be done centrally through a computer-generated randomisation sequence. One arm will be started on a prednisolone dose of 40mg/day for 7 days, followed by a placebo from day 8 to day 28 if Lille on Day 7 is < 0.45. The second arm will be started on prednisolone - 40mg per day for 7 days, followed by same dose for next 7 days if Lille is less than < 0.45. Lille scores will be calculated on Day 7; non-responders will discontinue the treatment. Patients will be screened for infections till 90 days from the day of initiation of prednisolone. The three patient arms will be compared for severity scores of the disease, rate and severity of infections, diabetic control, post treatment outcomes, and mortality. Patients enrolled in the study should not receive pentoxifylline, NAC, omega 3 fatty acid lipid emulsions, prophylactic antibiotics, granulocyte colony-stimulating factor, faecal microbiota transplantation or any other experimental therapies.

Sample size-A recent study (STASH) reported that 33.1% of patients with 28 day fixed dose steroid develop infections, and the investigators believe that 7 day steroid therapy may reduce infections significantly by 20% (13.1%) and with a power of 80%, significance level of 5%, the current study will need to include 66 in each arm, i.e., 132 in total. Considering a 10% attrition rate, the number of participants needed to included are 146 participants, i.e., 73 in each arm. Randomization will be done centrally at the primary centre, i.e., AIG Hospitals, by the clinical trial coordinators with a block size of 10 and randomized equally in a 1:1 ratio to either a 7-day steroid or 14-day steroid. Each center shall provide the details of respective CTCs or an individual who will contact the primary center CTC (at least 12 hours prior to the planned prednisolone initiation) for the randomized group.

STATISTICAL ANALYSIS - All patients who receive at least one dose of corticosteroids will be included in the analysis and performed intention-to-treat analysis. Descriptive statistics such as age, history of last alcohol intake, amount of alcohol, laboratory parameters (complete hemogram, liver function tests, renal function tests, procalcitonin levels) and severity scores will be expressed as mean with standard deviation (SD) for parametric data and median with interquartile range (IQR) for non-parametric continuous data if the data is skewed. Categorical data which include gender distribution, comorbidities, decompensations, use of drugs for treating patients, and each adverse events will be expressed as numbers (n, %) i.e., as proportions. Student's t-test will be used to compare continuous data between the two groups or Mann-Whitney U test for non-parametric data. Pearson's Chi-square test or two sided Fisher's exact test (when the observations are less than five) to compare categorical data between the three groups. The main outcomes will be reported as estimated effect sizes along with precision (95% confidence intervals [CIs]). Kaplan Meier survival analysis will be carried out to assess the incidence of infections and effect on survival at days 30 and 90. A preplanned sub-group analysis as required based on prednisolone response will be performed. A competing risk analysis will be performed, considering death and transplantation as competing events for infection. Using the Fine and Gray model to estimate the risk of infection on day 90, accounting for competing events, i.e., death or transplant. The time to event will be defined as the number of days from the initiation of prednisolone to the occurrence of infection, death or transplant, and the subdistribution hazard ratio (sHR) with the corresponding 95% CI will be calculated. Covariates with P<0.05 in the univariate analysis will be included in a multivariate model to identify independent predictors of infection. Statistical significance will be set at P < 0.05. All statistical tests were performed using SPSS and STATA as required.

AAH: AAH will be defined as per National Institute on Alcohol Abuse and Alcoholism (NIAAA) as the onset of jaundice (serum bilirubin >3 mg/dl) within two months of the last significant alcohol use, with aspartate aminotransferase >50 U/L and <400 U/L, aspartate aminotransferase/alanine aminotransferase ratio >1.5, and exclusion of other causes of liver disease in a patient with daily harmful alcohol use for ≥6 months.1 Biopsy will be performed in selected cases when the diagnosis is in question, and the patient is deemed fit enough to tolerate the invasive procedure.

Responder: A Lille score of <0.45 on day seven is considered as a responder to prednisolone.10 Patients with Lille's score ³0.45 are non-responders and should not continue prednisolone. Acute kidney injury: Increase in serum creatinine by ≥0.3 mg/dL within 48 h or a percentage increase serum creatinine ≥50% from baseline which is known, or presumed, to have occurred within the prior 7 days.11: Patients with diabetes mellitus, HbA1c >9, are considered uncontrolled diabetics and should not be included. Steroid withdrawal was identified by the presence of anorexia, fever, nausea, lethargy, malaise, arthralgias, desquamation of the skin, weakness, and weight loss occurring in varying combinations after stopping prednisolone.12 Patients with glomerular filtration rate < 60 ml/m/1.73m2 for three months will be considered as chronic kidney disease (CKD) and must not be included. Patients with acute variceal bleeding (within 7 days of the episode) shall not be included for at least 7 days (due to the risk of post-endotherapy-related ulcer bleeding with prednisolone). In rare instances, if the investigator desires to include patients with AVB before 7 days of the episode, documented evidence of healing on endoscopy is recommended. Patients with active uncontrolled infection (defined as persistent fever, leucocytosis, elevated procalcitonin [> one ng/ml], microbiologically proven infections or active signs of infection as shown in Table 2 below) will not be included. Such patients may be included once the infection is controlled for at least 48 hours and the cultures are sterile. All infections will be adjudicated and treated by the ID specialist blindly. At every visit, the patient meets the ID specialist.

Spontaneous bacterial peritonitis (SBP)-Ascitic fluid analysis done under strict aseptic precautions showing high serum albumin ascites gradient (SAAG), a low protein with a polymorphonuclear cell count of ≥250/mm3. Or patients with ascitic fluid gram stain/ culture positive

Secondary peritonitis- Neutrophil count ≥ 250/mm³ in ascitic fluid and evidence (abdominal CT/ surgery) of an intra-abdominal source of infection.

Urinary tract infection (UTI)-Uncomplicated urinary tract infection: At least 1 symptom of acute lower UTI (dysuria, urgency, frequency, or suprapubic tenderness) and a urine dipstick test result positive for either nitrites or leukocyte esterase.

1. Complicated Urinary tract infection: as having at least 2 of the following clinical criteria:

1. (1) chills, rigors, or fever (temperature ≥38.0°C);
2. (2) elevated white blood cell count (>10 000/mm3) or left shift (>15% immature polymorphonuclear leukocytes);
3. (3) nausea or vomiting;
4. (4) dysuria, increased urinary frequency, or urinary urgency; or
5. (5) lower abdominal pain or pelvic pain;

AND the presence of pyuria as evidenced by 1 of the following:

A. White blood cell count 10 cells/μL or greater in unspun urine; B. 10 or more cells per high-power field in urine sediment; or C. Positive leukocyte esterase on urinalysis; AND at least 1 associated risk factor, including indwelling catheter, neurogenic bladder, obstructive uropathy, azotemia due to renal disease, or urinary retention in men due to benign prostatic hypertrophy. Indwelling urinary catheters or devices (including nephrostomy tubes, indwelling stents, or both) were removed or replaced (if feasible) within 12 hours of randomization. Signs or symptoms of acute pyelonephritis could also be defined by flank pain or costovertebral angle tenderness on physical examination.

Pneumonia- 1. New pulmonary infiltrate in the presence of

1. At least one respiratory symptom (cough, sputum production, dyspnea or pleuritic pain) with
2. At least one finding on auscultation (rhonchi or creps) Or One sign of infection (core body temperature > 38 C or < 36 C or TLC (Total Leukocyte Count) > 10,000 or <4000/cu mm.

Cellulitis (skin and soft tissue infections)-Local warmth, tenderness, or acute pain; unilateral erythema or bilateral erythema, with a temporal association between symptoms and the more severely affected leg; and unilateral edema.

Spontaneous bacteremia (SB) - Positive blood cultures and no evident cause of bacteremia Secondary bacteremia - (1) catheter-related infection (positive blood and catheter cultures); (2) bacteremia occurring within 24 hours after an invasive procedure. Clostridium difficile infection (CDI)- Patients with unexplained and new-onset ≥3 unformed stools in 24 hours and the presence of C. difficile toxin A and B, or B alone, in stools as detected by EIA or NAAT.

CNS infection- Patients with symptoms and signs of meningitis and/or CSF analysis suggestive of infection.

Bone and joint infections 1. A clinical syndrome comprising any of the following; a) localized pain OR b) localized erythema OR c) temperature >38.0ºC OR d) a discharging sinus or wound.

a. Has a bone and joint infection in one of the following categories; a) Native osteomyelitis (i.e., bone infection without metalwork) including haematogenous or contiguous osteomyelitis, and long bone, skull, foot or other foci OR b) Native joint sepsis treated by excision arthroplasty OR c) Prosthetic joint infection treated by debridement and retention, by one stage revision or by excision of the prosthetic joint (with or without planned re-implantation) OR d) Orthopaedic device or bone-graft infection treated by debridement and retention, or by debridement and removal OR e) Spinal infection including discitis, osteomyelitis and/or epidural abscess.

Bacterial meningitis-

1.clinical presentation strongly suggestive of CABM, including signs such as neck stiffness, petechiae, headache, fever, confusion, or impaired level of consciousness, and at least one of the following:

1. Positive CSF culture
2. Positive blood culture and more than >10 leukocytes × 106/L in the CSF
3. Presence of bacteria in Gram stain of CSF Non-culture detection of bacteria in CSF by either bacterial antigen test or 16S rRNA gene amplification.

Fungal infections-

1. Candidiasis- Screening for oral candidiasis (Visual diagnosis)
2. If having non resolving fever with appropriate antibiotics - if invasive lines insitu/TPN/Abdomen surgery- candidiasis to be considered - culture and Beta D glucan for diagnosis
3. Invasive Pulmonology Aspergillus- Respiratory symptoms with CT suggestive of Nodules or GGO - Bronchoscopy BAL galactomannan +/- culture positive for Aspergillus - Diagnostic
4. Mucormycosis - Nasal/orbital symptoms - Tissue KOH broad aseptate hyphae - confirmed mucor
5. Cutaneous fungal infection - Tinea - clinical diagnosis
6. Fungal esophagitis- Demonstration of whitish plaques on endoscopy and smear Unknown source-the presence of fever, leucocytosis and tachycardia (requiring antibiotic therapy without any identifiable source.)

ELIGIBILITY:
Inclusion Criteria:

* Patients with AAH aged between 18 and 80 years with a MELD score >21 and/or mDF >32 will be included.
* Patients with infection at baseline will be included if they have controlled infection defined as afebrile for at least 48 hours, sterile cultures and procalcitonin < 1 ng/ml.

Exclusion Criteria:

* Age < 18 years, > 80 years
* Active Infection
* Persistent acute kidney injury (creatinine >1.5 mg/dl) or chronic kidney disease
* Recent/ongoing bleed
* Active peptic ulcer disease
* Hepatocellular carcinoma, portal vein thrombosis or hepatic venous outflow tract obstruction
* Patients with concomitant other liver diseases including hepatitis B, C
* Patients with HIV
* Uncontrolled diabetes mellitus
* Patients on pentoxifylline or NAC
* Patients who are unwilling

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-04-08 (Estimated); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants developing infection in each group | at day 28 and 90
  Infections will be assessed as defined priori. Infections will be compared among patient who respond to steroids and who do not.

SECONDARY OUTCOMES:
Mortality rate among the two groups | day 90
  Proportion of patients dying within the specified time period
Effiacy of prednisolone in each group | day 28 and 90
  Defined as proportion of patients achieving model for end-stage liver disease (MELD) score < 17. The minimum value of MELD is 6 and maximum is 40.
Number of steroid responders in each group | day 7
  response to prednisolone defined as Lille's <0.45
compare proportion of patients requiring readmission | day 90
  readmission in each group at day 90
compare incidence of acute kidney injury (AKI) In each group | day 90
  Acute kidney injury (AKI) will be defined as per the latest guidelines of International Ascites Club as an increase in serum creatinine ≥0.3 mg/dl (26.5 μmol/L) within 48 h or ≥50% from baseline value known or presumed to have occurred within the prior 7 days and/or urine output ≤0.5 ml/kg for ≥6 h
compare adverse events | day 90

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - AIG Hospitals, Hyderabad, Telangana
  - AIG, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: Yes
Infection data, mortality and outcomes as specified in the trial will be shared
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 1.1.2027 to 1.1.2029
Access Criteria: By mailing the specified protocol and ethics approval, any scientist can access the data by mailing to the primary investigator